CLINICAL TRIAL: NCT05812794
Title: TOlerability of Transcranial Direct Current Stimulation in Pediatric Stroke Survivors
Acronym: TOPSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Stuart Mason Fraser, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0092
Record Dates: First submitted 2023-03-30; First posted 2023-04-14 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-08

CONDITIONS: Childhood Stroke
Keywords: neuromodulation; transcranial direct current stimulation; stroke; rehabilitation; childhood stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Transcranial Direct Current Stimulation (tDCS) (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Participants will come for 5 sequential days of 2 hour long occupational therapy sessions augmented by tDCS for the first 20 minutes of the session. At arrival, the "stimulation safety sheet" will be completed by the occupational therapist.The saline soaked electrodes will be placed on the study subjects head and connected to the Soterix 1x1 Limited Total Energy (LTE) enabled tDCS device. Current output through the device will be sham stimulation on day 1 , followed by steady increases to a maximum of 1milliampere (mA) in patients aged 5-12 years old, and 1.5 mA in patients aged 13-19 years old, per the study design flow sheet at the end of this protocol. Blood pressure, pulse rate, and peg-board scores will be recorded as indicated on the stimulation safety sheet during each session.A repeat assessment will be done by the occupational therapist one week post therapy completion.There will be a repeat assessment visit 3 months post intervention.

SUMMARY:
The purpose of this study is to evaluate the tolerability of tDCS in childhood stroke survivors and to assess for improvement in arm function in patients receiving tDCS and occupational therapy

ELIGIBILITY:
Inclusion Criteria:

* Childhood stroke survivor - either arterial ischemic stroke or intracerebral hemorrhage.
* Stroke must be childhood onset, defined as occurring day 29 of life to 18 years of age (per the American Heart Association's definition of childhood stroke)
* 3 months or greater from stroke onset
* Arm impairment, defined as pediatric stroke outcome measure of 1 or greater of affected arm.
* Affected arm Fugl-Meyer score of 60 or lower.
* Able to participate in occupational therapy sessions.

Exclusion Criteria:

* Uncontrolled epilepsy, defined as seizure within the past 6 months.
* Craniectomy without replacement of bone flap. Patients who underwent craniectomy will need the bone flap reattached prior to participation.
* Presence of cranial metal implants or implant device that could be affected by tDCS: cochlear implant, implanted brain stimulator, or programmable ventriculoperitoneal shunt.

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Fraser, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fraser S, Clearman A, Abrahams M, Gillick B, Lal T, Savitz S, Yozbatiran N. TOPSS: TOlerability of transcranial direct current stimulation in Pediatric Stroke Survivors. Front Hum Neurosci. 2025 Aug 5;19:1629499. doi: 10.3389/fnhum.2025.1629499. eCollection 2025. PMID 40836943

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 15 [6 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5
Age at stroke [Mean (Standard Deviation); unit: years] | 10.1 (7.14)
Type of Stroke [Count of Participants; unit: Participants]
  Intracranial Hemorrhage | 2
  Arterial Ischemic | 3
Arm affected [Count of Participants; unit: Participants]
  left arm affected | 3
  right arm affected | 2
Number of participants with history of seizures at stroke presentation [Count of Participants; unit: Participants] | 4
Number of participants with a diagnosis of epilepsy [Count of Participants; unit: Participants] | 2
Number of prescribed antiepileptics [Mean (Standard Deviation); unit: Number of prescribed antiepileptics] | 1 (1.22)
Global Function as Assessed by Score on the Pediatric Stroke Outcome Measure (PSOM) Rating Scale [Median (Full Range); unit: score on a scale] — The Pediatric Stroke Outcome Measure is a physician-administered rating scale of global function scored from 0 (no deficit) to 10 (profound deficit, immobile and non-responsive). Total score ranges from 0 to 10, with a higher score indicating a greater deficit in function.
  score on a scale | 2 [1 to 4]
Stroke Etiology [Count of Participants; unit: Participants]
  Aneurysm Rupture | 1
  Traumatic Dissection | 1
  Meningitis and Disseminated Intravascular Coagulation | 1
  Focal Cerebral Arteriopathy | 1
  Complication of Cerebral Arteriovenous Malformation Embolization | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Complete the Study
Time Frame: 1-week post therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 5
Participants | 5

2. Primary Outcome: Arm Function as Assessed by the Fugl-Meyer Score of Upper Extremity Function
Description: Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform; 1=performs partially; and 2=performs fully. Total score ranges from 0 to 66, with a higher score indicating greater arm function.
Time Frame: 1 week post therapy
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 5
score on a scale | 41 [38 to 43]

3. Secondary Outcome: Tolerability as Assessed by the Number of Patients That Endorse Any Side Effects as Documented on the Stimulation Monitoring Sheet
Time Frame: immediately post stimulation Day 1, immediately post stimulation Day 2, immediately post stimulation Day 3, immediately post stimulation Day 4, immediately post stimulation Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 5
Participants
  immediately post stimulation Day 1 | 4
  immediately post stimulation Day 2 | 2
  immediately post stimulation Day 3 | 2
  immediately post stimulation Day 4 | 1
  immediately post stimulation Day 5 | 2

4. Secondary Outcome: Tolerability as Assessed by the Number of Patients With Hypotension or Hypertension on Blood Pressure Monitoring
Time Frame: From baseline to 1 week post-therapy session
Measure: Count of Participants; unit: Participants
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 5
Participants | 0

5. Secondary Outcome: Tolerability as Assessed by the Number of Patients With a Decrease in Score of 5 or Greater on the Peg-Board Test
Description: The peg-board test is scored from 0 to 50, with the score indicating the number of pegs placed correctly into the board using the affected hand. A higher score indicates a better outcome, and a decrease in score over time indicates worsening of functioning over time. The number of participants with a decrease in score of 5 or greater on the peg-board test is reported.
Time Frame: Baseline, immediately post stimulation Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 5
Participants | 0

6. Secondary Outcome: Arm Function as Assessed by the Fugl-Meyer Score of Upper Extremity Function
Description: as for outcome 2
Time Frame: 3 month post therapy
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 5
score on a scale | 42 [37 to 44]

7. Secondary Outcome: Change in Quality of Unilateral Upper Limb Movement as Assessed by the Melbourne Assessment of the Upper Extremity (MUUL)
Description: This assessment has a total score range of 0-100% a higher score indicating better outcome
Time Frame: Baseline,1 week post therapy , 3 months post therapy
Population: Data were not collected for this outcome measure.
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Global Function as Assessed by Score on the Pediatric Stroke Outcome Measure (PSOM) Rating Scale
Description: The Pediatric Stroke Outcome Measure is a physician-administered rating scale of global function scored from 0 (no deficit) to 10 (profound deficit, immobile and non-responsive). Total score ranges from 0 to 10, with a higher score indicating a greater deficit in function.
Time Frame: 1 week post therapy
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 5
score on a scale | 2 [1 to 4]

9. Other Pre Specified Outcome: Global Function as Assessed by Score on the Pediatric Stroke Outcome Measure (PSOM) Rating Scale
Description: as for outcome 8
Time Frame: 3 months post therapy
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 5
score on a scale | 2 [1 to 4]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Transcranial Direct Current Stimulation (tDCS)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transcranial Direct Current Stimulation (tDCS) (N=5)
Itchiness (General disorders) | 5
Tingling (General disorders) | 2
Unusual feelings on skin of head (General disorders) | 1
Sleepiness (General disorders) | 2
Change in hearing (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT05812794/Prot_SAP_000.pdf